CLINICAL TRIAL: NCT06412562
Title: The Maudsley 3-item Visual Analogue Scale (M3VAS) Validation in Polish Population Diagnosed With Major Depressive Episode
Brief Title: M3VAS Validation in Polish Population
Status: Recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: M3VAS_PL
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Depressive Disorder
Keywords: anhedonia; low mood; suicidality; depression; m3vas
MeSH Terms: conditions — Depressive Disorder; Anhedonia; Consciousness Disorders; Suicidal Ideation; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major Depressive Episode: Patients must have a Diagnostic and Statistical Manual 5 (DSM-5) diagnosis of Major Depressive Disorder (MDD) or Bipolar Disorder (BD), as determined by a psychiatrist.
  Interventions: Diagnostic Test: The Maudsley 3-item Visual Analogue Scale (M3VAS)

INTERVENTIONS:
Diagnostic Test: The Maudsley 3-item Visual Analogue Scale (M3VAS) — Patients will be asked to complete The Maudsley 3-item Visual Analogue Scale (M3VAS) and 16-item Quick Inventory of Depressive Symptomatology (QIDS-SR-16).
  Other Names: 16-item Quick Inventory of Depressive Symptomatology (QIDS-SR-16)

SUMMARY:
Low mood and anhedonia represent the fundamental symptoms of major depressive disorder (MDD). Nevertheless, there is currently no standardized visual analogue scale available to assess the extent of both symptoms concurrently. The Maudsley 3-item Visual Analogue Scale (M3VAS) is a newly developed tool for participants to self-assess core symptoms of depression: mood quality, pleasure experience (anhedonia), and suicidality. Despite suicidality not being a primary symptom, it is included due to its critical relevance to safety. Participants will be instructed to rate the intensity and frequency of their experiences over the preceding two weeks by marking a 100 mm ungraded line. A researcher will then assign a numerical value based on the mark's position, utilizing the left edge as 0 and the right as 100. The total score range, combining the three symptoms, ranged from 0 (minimum) to 300 (maximum). The M3VAS exhibited good psychometric properties in British population. In this study, the objective is to assess the psychometric properties of the scale within the Polish population diagnosed with major depressive episode within major depressive disorder or bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis as provided by DSM-5 criteria:

Major depressive disorder (MDD) Bipolar disorder (BD)

Exclusion Criteria:

Diagnosis as provided by DSM-5 criteria:

Psychotic disorders Current Mania or hypomania within bipolar disorder (BD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients referred to the tertiary-reference unit for mood disorders with MDD or BD diagnosis, currently either with current depression or euthymic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The Maudsley 3-item Visual Analogue Scale (M3VAS) | Baseline
  To analyze internal consistency and factor analysis

SECONDARY OUTCOMES:
16-item Quick Inventory of Depressive Symptomatology (QIDS-SR-16) | Baseline
  To analyze convergent validity with The Maudsley 3-item Visual Analogue Scale (M3VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moulton CD, Strawbridge R, Tsapekos D, Oprea E, Carter B, Hayes C, Cleare AJ, Marwood L, Mantingh T, Young AH. The Maudsley 3-item Visual Analogue Scale (M3VAS): Validation of a scale measuring core symptoms of depression. J Affect Disord. 2021 Mar 1;282:280-283. doi: 10.1016/j.jad.2020.12.185. Epub 2020 Dec 31. PMID 33418379